CLINICAL TRIAL: NCT00682526
Title: Pre-hospital Wireless Transmission of Electrocardiograms to a Cardiologist Via a Hand-held Device: The TIME Multicenter Study
Brief Title: Pre-Hospital Wireless Transmission of Electrocardiograms to a Cardiologist Via a Hand-Held Device
Status: Completed | Type: Observational
Sponsor: Welch Allyn (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: TIME Multicenter Study
Record Dates: First submitted 2008-05-12; First posted 2008-05-22 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Myocardial Infarction
Keywords: EMS patients with intention to treat with coronary reperfusion therapy (PCI or thrombolytics) based on their initial presentation
MeSH Terms: conditions — Myocardial Infarction | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pre-study Period (Group 1 and Group 2).: The TIME-MC study was conducted from June 2003 to June 2008 at NEMC (Figure 1) and from May 2005 to September 2008 at the six larger medical centers (Figure 2). Two groups were studied. Group 1 included patients at NEMC and Group 2 included patients at the other six medical sites. The study was divided into three periods:
  Pre-study period (Group 1 and Group 2). No PH-ECG transmission system was available.
- Study Period (Group 1 and Group 2): Study period (Group 1 and Group 2). PH-ECG transmission to a cardiologist's hand-held device was attempted through pre-assigned EMS ambulances equipped with a wireless ECG transmission device in addition to a STEMI code system. In Group 1, this referred to the pilot study at NEMC from June 2003 to May 2005.
  Interventions: Device: SmartLink Wireless Monitoring System (K033642)
- Post-study period (Group 1): Post-study period (Group 1). PH-ECG transmission and a STEMI code system implemented after the pilot study period.
  Interventions: Device: SmartLink Wireless Monitoring System (K033642)

INTERVENTIONS:
Device: SmartLink Wireless Monitoring System (K033642) — All EMS transported patients age 18 or over who have their ECG attempted to be wirelessly transmitted and with the intention to treat with coronary reperfusion therapy (PCI or thrombolytics)based on their initial presentation.
  Other Names: Wireless transmission of ECG with intention to treat with coronary reperfusion therapy.
  Groups: Post-study period (Group 1); Study Period (Group 1 and Group 2)

SUMMARY:
Aim: To determine the impact of wireless transmission of prehospital ECGs to a hand-held computer on time to treatment and myocardial salvage in acute MI patients.

Background: The TIME-1 investigators documented a 27% (109 to 80 minutes) reduction of time from EMT arrival at the scene to successful primary PCI implementing pre-hospital ECG transmission to the ED. ECG transmission directly to a physician's cellular phone/PDA through a wireless modem has only recently become an option. The recently completed TIME-NorthEast (NE) study tested the Welch Allyn version of this system and the results show a reduction in time to reperfusion for acute MI patients by 66 minutes (116 to 50).

Methods: This study will involve approximately 20 sites around the country. The study will be divided into two phases: a consecutive control data collection phase (Phase I) and an intervention with concurrent control phase (Phase II). Phase II will begin after installation of Welch Allyn ECG transmission equipment. The primary end-point will be time to reperfusion and secondary end-points will include myocardial salvage, aborted infarction and hospital mortality. ECG measurements will be made at a central ECG core lab by a blinded investigator.

Data Analysis: Patient characteristics for the three periods were compared with the chi-square statistic for categorical variables and one-way analysis of variance for age. The Wilcoxon rank-sum statistic was used to compare time-to-reperfusion in the pre-study and study periods as well as in the Group 1 post-study period. Comparisons were performed separately for EMS and self-transport groups.

ELIGIBILITY:
Inclusion Criteria:

All patients with a diagnosis of acute STEMI defined as 1 mm ST segment elevation in two spatially contiguous leads were included. There were two major subgroups: emergency medical services (EMS) and self-transport patients. Self-transport patients, who did not have PH-ECG transmission, served as a comparison group.

Exclusion Criteria:

* Less than age 18
* No intent to undergo reperfusion therapy (PCI or thrombolytics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: EMS transported patients age 18 or over who have their ECG attempted to be wirelessly transmitted and with the intention to treat with coronary reperfusion therapy (PCI or thrombolytics) based on their initial presentation All self transported and EMS transported patients age 18 or over with the intention to undergo reperfusion therapy (PCI or thrombolytics)based on their initial presentation who do not qualify for the intervention group.
Sampling Method: Non-Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2003-06; Primary Completion 2008-09 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Door to intervention time - time from emergency department door time until intervention. | time from emergency department door time until intervention.

SECONDARY OUTCOMES:
Salvaged myocardial tissue - pre-hospital ECGs will be read using the Aldrich final MI size prediction to calculate the size of infarct that would be expected to result without reperfusion treatment. | pre hospital ECG - discharge ECG
Aborted infarction-defined as combined ECG and cardiac biomarkers criteria:1.subsiding of ST deviation greater than or equal to 50% within 2 hours after reperfusion treatment. 2.rise in cardiac enzymes less than or equal to 2 times upper value of normal. | 2 hours after reperfusion treatment
Hospital mortality - whether the patient was discharged alive. | discharge
No infarct related artery at time of heart catheterization. | catheterization

CONTACTS AND LOCATIONS:
Overall Officials: Galen S Wagner, MD, Principal Investigator — Duke University
Locations (7):
- United States (7):
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - Shands @ AGH, Gainesville, Florida
  - South Miami Heart Center, Miami, Florida
  - Durham Regional Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Bethesda North Hospital, Cincinnati, Ohio
  - University of Pittsburgh Medical Center - Presbyterian, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Adams G, Abusaid G, Lee B, Maynard C, Campbell P, Wagner G, Barbagelata A. From theory to practice: implementation of pre-hospital electrocardiogram transmission in ST-elevation myocardial infarction - a multicenter experience. J Invasive Cardiol. 2010 Nov;22(11):520-5. PMID 21041847